CLINICAL TRIAL: NCT05055219
Title: Conventional and Metabolomic Predictors of Prediabetes & Insulin Resistance
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Joyce Lee, MD, MPH, University of Michigan
Other Study IDs: HUM00006955; 5R01HD074559-05 (NIH)
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: PreDiabetes; Obesity, Childhood
MeSH Terms: conditions — Prediabetic State; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Overweight or Obese Group (visits #1-4): Children and young adults who are 8 to 22 years of age, who have risk factors for diabetes such as being overweight. Overweight or obese, as defined by a BMI ≥ 85th percentile & <95th percentile or BMI ≥ 95th percentile, respectively. Study participants cannot be pregnant or currently take medications known to affect glucose metabolism including, metformin, oral steroids, sulfonylureas, and insulin.
- Group 2: Overweight or Obese Group (visits #3-4): Children and young adults who are 8 to 22 years of age, who have risk factors for diabetes such as being overweight, or children and young adults who previously participated in the study (completed visits #1-2 in previous study phase). Overweight or obese, as defined by a BMI ≥ 85th percentile & <95th percentile or BMI ≥ 95th percentile, respectively. Study participants cannot be pregnant or currently take medications known to affect glucose metabolism including, metformin, oral steroids, sulfonylureas, and insulin.
- Group 3: Normal Weight Control Group: Children and adolescents who are 8 to 17 years of age, who have do not have risk factors for diabetes such as being overweight or a history of type 2 diabetes in the family. Healthy weight, as defined by a BMI ≥ 5th percentile & < 85th percentile. Study participants cannot be pregnant or currently take medications known to affect glucose metabolism including, metformin, oral steroids, sulfonylureas, and insulin.

SUMMARY:
The purpose of this study is to evaluate the longitudinal test performance of an array of conventional biomarkers of glycemia, including Hemoglobin A1c (HbA1c), and novel metabolomic biomarkers for identifying progression of glucose tolerance (normal to prediabetes or prediabetes to diabetes) in an overweight and obese pediatric cohort.

ELIGIBILITY:
Inclusion Criteria:

* Groups 1 and 2 (overweight and obese groups):
* Age 8-17 years for the visits #1 and #2, individuals can be as old as 22 years for follow-up visits #3 and 4
* Overweight or obese, as defined by a BMI ≥ 85th% & <95th% or BMI ≥ 95th%, respectively by age and sex, and for those 16 years and older, BMI ≥25 and <30 and BMI ≥30
* For Group 2 only: previously completed visits 1-2 in 2007-2013 and formally agreed to be re-contacted for study purposes
* Group 3 (Normal weight controls):
* Age 8-17 years
* Healthy weight, as defined by a BMI ≥ 5th percentile & < 85th percentile, respectively by age and sex

Exclusion Criteria:

* Previous diagnosis of type 1 diabetes
* Use of concurrent medications known to affect glucose metabolism (metformin, oral steroids, sulfonylureas, insulin)
* Verbal report of Pregnancy

Ages: 8 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will consist of normal weight, overweight or obese individuals aged 8 to 17 years at visits #1 and #2, and can be as old as 22 years for follow-up visits #3 and #4. Participants will be recruited from a variety of sites including University Michigan clinical sites, non-University of Michigan clinical sites, schools in the local area, and the University Michigan medical school campus. Participants from Group 2 (visits #3-4) completed visits #1-2 in 2007-2013 and formally agreed to be re-contacted for study purposes.
Sampling Method: Non-Probability Sample
Enrollment: 772 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Progression of glucose tolerance | Up to 5 years
  Normal glucose tolerance, prediabetes, or diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Lee, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States